CLINICAL TRIAL: NCT04749888
Title: Impact of the Korea Early Childhood Home-visiting Intervention on Childhood Health and Development and Maternal Health: A Randomized Controlled Community Trial
Brief Title: Impact of the Korea Early Childhood Home-visiting Intervention
Acronym: KECHI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government); Seoul National University (Other); Hanyang University (Other); Soon Chun Hyang University (Other); Kangwon National University (Other); University of Ulsan (Other)
Responsible Party: Principal Investigator, Young-Ho Khang, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C-1911-150-1083; HI19C0481, HC19C0048 (Other Grant/Funding Number: Ministry of Health and Welfare, Republic of Korea); RS-2025-00516414 (Other Grant/Funding Number: National Research Foundation of Korea); KCT0005579 (Registry Identifier: World Health Organization [WHO] Registry Network)
Record Dates: First submitted 2020-11-05; First posted 2021-02-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Child Development; Parenting; Infant Development; Pregnancy Related; Maternal Distress
Keywords: Home visiting; Child health and development; Maternal health; Randomized controlled trial; Community intervention trial; Nurse home visiting; Republic of Korea; Prenatal and early childhood periods

STUDY DESIGN:
Masking Description: The research management staff, home visit nurses (intervention teams), and study participants will be aware of the allocation results. However, the research nurses making outcome assessments will be blinded to the randomization, and families will be asked not to disclose their group status during the surveys. The research nurses (outcome assessors) will only be notified of the survey schedules (6 weeks, 6 months, 12 months, and 24 months) of both groups so that the outcome indicators can be measured with blinding maintained. Statistical analysts will not be able to access the randomization variable until all 2 years of data are collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Targeted nurse-led home visiting (Experimental): The intervention group will receive 25-29 home visits during pregnancy and the first 2 years of life conducted by child health nurses. The frequency of home visits will be determined by nurses based on the needs of the families. The content of each home visit is individually tailored to the mother's needs, skills, strengths, and capacity using parenting education materials.
  Interventions: Behavioral: Targeted nurse-led home visiting
- Control group (No Intervention): The control group will receive existing maternal and child health services (usual care) except for the targeted nurse-led home visits.

INTERVENTIONS:
Behavioral: Targeted nurse-led home visiting — The KECHI encompasses 25-29 home visits, group activities, and community service linkage by social workers from the prenatal period until the child reaches the age of 2 years; as such, it is a complex intervention involving various domains to address a wide range of outcomes. Pregnant women with two or more risk factors who are deemed to have difficulties in raising children are eligible for the targeted multiple nurse home visits. Each home visit is implemented based on families' needs, and individualized interventions are provided to improve parenting and the home environment in order to promote the child's health and development and maternal health. The program includes educational materials for parents, such as a booklet covering issues on prenatal care, child development, postnatal child care, parent-child attachment, play, communication, safety, and goal-setting.
  Other Names: KECHI (Korea Early Childhood Home-visiting Intervention)
  Arms: Targeted nurse-led home visiting

SUMMARY:
Maternal and early childhood home visits have been proposed as an effective strategy to improve the health and development of disadvantaged children. In South Korea (hereafter, Korea), a maternal and early childhood home visit program has been implemented since 2013 in Seoul, and then was adopted in 2019 by the central government as a national policy for child health and development.

The Korea Early Childhood Home-visiting Intervention (KECHI) encompasses 25-29 home visits, group activities, and community service linkage by social workers from the prenatal period until the child reaches the age of 2 years; as such, it is a complex intervention involving various domains to address a wide range of outcomes. Each home visit is implemented based on the family's needs, and individualized interventions are provided to improve parenting and the home environment in order to promote children's health and development and maternal health.

This study is a randomized controlled community trial conducted in Korea to examine the impact of targeted home visits led by nurses in the prenatal and early childhood period on children's health and development and maternal health.

This study is a superiority trial with two parallel groups from pregnancy until the child reaches 2 years of age. Pregnant women with two or more risk factors will be recruited to participate in the study after they provide informed consent. Participants will then be randomly assigned to the intervention or control group with a 1:1 allocation through an independent web-based random allocation system. We expect a total of 800 families (400 families in each group) to be recruited. The intervention group will receive the KECHI program and the control group will receive existing maternal and child health services (usual care), but not multiple home visits by nurses. Both groups will receive gift cards of 30,000 Korean won (about 27 USD) for each round of surveys.

The intervention and control groups will be surveyed on the outcome variables of home environment, child development, breastfeeding, maternal health, child hospital visits due to injuries, and community service linkage at four home visits by trained research nurses at baseline and at 6 months, 12 months, and 24 months after birth. Telephone contact will also be made at 6 weeks and 18 months after birth for both groups. Outcome measurements will be performed by research nurses and data management will be conducted by statistical analysts. The analysis will be conducted for the intention-to-treat (ITT) and per-protocol (PP) groups, with an interim analysis of outcomes up to the 6-month follow-up. For the primary outcomes and certain secondary outcomes, subgroup analyses will be performed based on factors such as region, fertility status, number of risk factors, presence of depression, education level, etc. Furthermore, this study will utilize administrative data available for all study participants to evaluate both short and long-term impacts of the KECHI intervention on maternal and child outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with two or more risk factors at the time of screening
* Pregnant women at less than 37 weeks of gestation
* Pregnant women who can read and answer questionnaires in Korean

Exclusion Criteria:

* Pregnant women who have experienced any critical event such as termination of pregnancy, stillbirth, or child death
* Pregnant women who plan to move abroad or to other regions where the KECHI service is not available within the next 6 months

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2045-12-31 (Estimated)

PRIMARY OUTCOMES:
Home environment | when the child is 6 months old.
  Home environment as assessed using IT-HOME (Infant-Toddler Home Observation for Measurement of Environment) when the child is 6 months old. IT-HOME (Infant-Toddler Home Observation for Measurement of Environment), composed of 45 items, was developed by Caldwell & Bradley (1984). The minimum score is 0 and the maximum score is 45, and a higher score means a better outcome.
Home environment | when the child is 12 months old.
  Home environment as assessed using IT-HOME (Infant-Toddler Home Observation for Measurement of Environment) when the child is 12 months old. IT-HOME (Infant-Toddler Home Observation for Measurement of Environment), composed of 45 items, was developed by Caldwell & Bradley (1984). The minimum score is 0 and the maximum score is 45, and a higher score means a better outcome.
Home environment | when the child is 24 months old.
  Home environment as assessed using IT-HOME (Infant-Toddler Home Observation for Measurement of Environment) when the child is 24 months old. IT-HOME (Infant-Toddler Home Observation for Measurement of Environment), composed of 45 items, was developed by Caldwell & Bradley (1984). The minimum score is 0 and the maximum score is 45, and a higher score means a better outcome.
Emergency department visits due to injuries | when the child is 6 weeks old.
  Number of emergency department visits due to injuries when the child is 6 weeks old.
Emergency department visits due to injuries | when the child is 6 months old.
  Number of emergency department visits due to injuries when the child is 6 months old.
Emergency department visits due to injuries | when the child is 12 months old.
  Number of emergency department visits due to injuries when the child is 12 months old.
Emergency department visits due to injuries | when the child is 24 months old.
  Number of emergency department visits due to injuries when the child is 24 months old.
Child development (K-Bayley-III) | when the child is 24 months old.
  Child development as assessed using the K-Bayley-III (Korean Bayley Scales of Infant and Toddler Development-III) score when the child is 24 months old
Breastfeeding duration | when the child is 6 weeks old.
  Breastfeeding duration when the child is 6 weeks old.
Breastfeeding duration | when the child is 6 months old.
  Breastfeeding duration when the child is 6 months old.
Breastfeeding duration | when the child is 12 months old.
  Maternal self-rated health when the child is 12 months old.
Breastfeeding duration | when the child is 24 months old.
  Breastfeeding duration when the child is 24 months old.
Maternal self-rated health | when the child is 6 weeks old.
  Maternal self-rated health when the child is 6 weeks old.
Maternal self-rated health | when the child is 6 months old.
  Maternal self-rated health when the child is 6 months old.
Maternal self-rated health | when the child is 12 months old.
  Maternal self-rated health when the child is 12 months old.
Maternal self-rated health | when the child is 18 months old.
  Maternal self-rated health when the child is 18 months old.
Maternal self-rated health | when the child is 24 months old.
  Maternal self-rated health when the child is 24 months old.
Community service linkage | when the child is 12 months old.
  Community service linkage as measured by the number of community services a mother has received during the last year when the child is 12 months old.
Community service linkage | when the child is 24 months old.
  Community service linkage as measured by the number of community services a mother has received during the last year when the child is 24 months old.
School readiness (EDI) | when the child is 66 months old
  School readiness as assessed using the Korean Early Development Instrument (EDI) administered by the child's teacher. The EDI evaluates children's overall developmental readiness for school across five domains: (1) Physical Health and Well-being, (2) Social Competence, (3) Emotional Maturity, (4) Language and Cognitive Development, and (5) Communication Skills and General Knowledge. The assessment consists of approximately 100 items based on teacher observations and takes 15-20 minutes per child to complete.
Child Intelligence (WPPSI) | when the child is 66 months old
  Child intelligence assessed using the Wechsler Preschool and Primary Scale of Intelligence (WPPSI-IV) administered by trained occupational therapist. The assessment measures overall intellectual ability and cognitive development.
Child abuse | when the child is 66 months old
  Number of child abuse reports obtained through secondary data linkage with the Social Security Information Service's child abuse reporting database.
Emergency department visits due to injuries (administrative data) | when the child is 66 months old
  Number of emergency department visits due to injuries (indirect indicator of child abuse) obtained via linkage with Korea National Health Insurance Service (NHIS) claims data.
Maternal depression (PHQ-9) | when the child is 42 months old
  Maternal depression as assessed using the PHQ-9 (Patient Health Questionnaire-9) when the child is 42 months old. The PHQ-9 (Patient Health Questionnaire-9) was developed by Kroenke, K. et al. (2001) as a tool measuring the depression level of adults and composed of 9 items. The minimum score is 0 and the maximum score is 27, and higher score means a worse outcome.
Maternal depression (PHQ-9) | when the child is 54 months old
  Maternal depression as assessed using the PHQ-9 (Patient Health Questionnaire-9) when the child is 54 months old. The PHQ-9 (Patient Health Questionnaire-9) was developed by Kroenke, K. et al. (2001) as a tool measuring the depression level of adults and composed of 9 items. The minimum score is 0 and the maximum score is 27, and higher score means a worse outcome.
Maternal depression (PHQ-9) | when the child is 66 months old
  Maternal depression as assessed using the PHQ-9 (Patient Health Questionnaire-9) when the child is 66 months old. The PHQ-9 (Patient Health Questionnaire-9) was developed by Kroenke, K. et al. (2001) as a tool measuring the depression level of adults and composed of 9 items. The minimum score is 0 and the maximum score is 27, and higher score means a worse outcome.
Maternal parenting behavior | when the child is 42 months old
  Maternal parenting behavior as assessed using a 17-item questionnaire measuring two dimensions: warm/responsive parenting and controlling parenting when the child is 42 months old. The warm/responsive dimension includes 9 items adapted by the Korea Institute of Child Care and Education from the Parental Style Questionnaire (Bornstein et al., 1996). The controlling dimension includes 8 items adapted by the Korea Institute of Child Care and Education based on Cho et al. (1999). Responses are rated on a 5-point Likert scale, with higher scores indicating greater endorsement of each parenting style.
Maternal parenting behavior | when the child is 54 months old
  Maternal parenting behavior as assessed using a 17-item questionnaire measuring two dimensions: warm/responsive parenting and controlling parenting when the child is 54 months old. The warm/responsive dimension includes 9 items adapted by the Korea Institute of Child Care and Education from the Parental Style Questionnaire (Bornstein et al., 1996). The controlling dimension includes 8 items adapted by the Korea Institute of Child Care and Education based on Cho et al. (1999). Responses are rated on a 5-point Likert scale, with higher scores indicating greater endorsement of each parenting style.
Maternal parenting behavior (32-PSDQ) | when the child is 66 months old
  Maternal parenting behavior as assessed using the 32-item Parenting Style and Dimensions Questionnaire (32-PSDQ), measuring authoritative, authoritarian, and permissive parenting styles, adapted from Robinson et al. (2001) and used in the Korean Early Childhood Education and Care Panel Study.
Cognitive-stimulating home environment (Parent-child interaction) | when the child is 42 months old
  Cognitive-stimulating home environment as assessed using the Home Environment Activities and Cognitive Stimulation (HEQ) questionnaire adapted from the Early Childhood Longitudinal Study Kindergarten Cohort (ECLS-K) when the child is 42 months old. The Korean version was translated by the Korea Institute of Child Care and Education. The instrument consists of 10 items measuring frequency of cognitive stimulation activities between parents and children over the past week, rated on a 4-point scale.
Cognitive-stimulating home environment (Parent-child interaction) | when the child is 54 months old
  Cognitive-stimulating home environment as assessed using the Home Environment Activities and Cognitive Stimulation (HEQ) questionnaire adapted from the Early Childhood Longitudinal Study Kindergarten Cohort (ECLS-K) when the child is 54 months old. The Korean version was translated by the Korea Institute of Child Care and Education. The instrument consists of 10 items measuring frequency of cognitive stimulation activities between parents and children over the past week, rated on a 4-point scale.
Cognitive-stimulating home environment (Parent-child interaction) | when the child is 66 months old
  Cognitive-stimulating home environment as assessed using the Home Environment Activities and Cognitive Stimulation (HEQ) questionnaire adapted from the Early Childhood Longitudinal Study Kindergarten Cohort (ECLS-K) when the child is 66 months old. The Korean version was translated by the Korea Institute of Child Care and Education. The instrument consists of 10 items measuring frequency of cognitive stimulation activities between parents and children over the past week, rated on a 4-point scale.

SECONDARY OUTCOMES:
Safety knowledge | when the child is 6 months old.
  Safety knowledge as measured by the number of questions the mother answered correctly about child accident prevention when the child is 6 months old. The questionnaire testing mothers' safety knowledge is composed of five items from the Korean National Health Insurance Service's Infant Health Examination Questionnaire.
Safety knowledge | when the child is 12 months old.
  Safety knowledge as measured by the number of questions the mother answered correctly about child accident prevention when the child is 12 months old. The questionnaire testing mothers' safety knowledge is composed of five items from the Korean National Health Insurance Service's Infant Health Examination Questionnaire.
Safety knowledge | when the child is 24 months old.
  Safety knowledge as measured by the number of questions the mother answered correctly about child accident prevention when the child is 24 months old. The questionnaire testing mothers' safety knowledge is composed of five items from the Korean National Health Insurance Service's Infant Health Examination Questionnaire.
Emergency department visits | when the child is 6 weeks old.
  Number of emergency department visits when the child is 6 weeks old.
Emergency department visits | when the child is 6 months old.
  Number of emergency department visits when the child is 6 months old.
Emergency department visits | when the child is 12 months old.
  Number of emergency department visits when the child is 12 months old.
Emergency department visits | when the child is 24 months old.
  Number of emergency department visits when the child is 24 months old.
Hospital admission | when the child is 6 weeks old.
  Number of hospital admission when the child is 6 weeks old.
Hospital admission | when the child is 6 months old.
  Number of hospital admission when the child is 6 months old.
Hospital admission | when the child is 12 months old.
  Number of hospital admission when the child is 12 months old.
Hospital admission | when the child is 24 months old.
  Number of hospital admission when the child is 24 months old.
Child development (Denver II) | when the child is 6 months old.
  Child development as assessed using Denver (Denver Developmental Screening Test) II when the child is 6 months old.
Child development (Denver II) | when the child is 12 months old.
  Child development as assessed using Denver (Denver Developmental Screening Test) II when the child is 12 months old.
Child development (Denver II) | when the child is 24 months old.
  Child development as assessed using Denver (Denver Developmental Screening Test) II when the child is 24 months old.
Premature birth | when the child is 6 weeks old.
  Premature birth as assessed by asking the mother whether the child was delivered before 37 weeks.
Delayed growth - height | when the child is 6 months old.
  Height in centimeters measured by a physical examination of the child when the child is 6 months old.
Delayed growth - height | when the child is 12 months old.
  Height in centimeters measured by a physical examination of the child when the child is 12 months old.
Delayed growth - height | when the child is 24 months old.
  Height in centimeters measured by a physical examination of the child when the child is 24 months old.
Delayed growth - weight | when the child is 6 months old.
  Weight in kilograms measured by a physical examination of the child when the child is 6 months old.
Delayed growth - weight | when the child is 12 months old.
  Weight in kilograms measured by a physical examination of the child when the child is 12 months old.
Delayed growth - weight | when the child is 24 months old.
  Weight in kilograms measured by a physical examination of the child when the child is 24 months old.
Delayed growth - head circumference | when the child is 6 months old.
  Head circumference in centimeters measured by a physical examination of the child when the child is 6 months old.
Delayed growth - head circumference | when the child is 12 months old.
  Head circumference in centimeters measured by a physical examination of the child when the child is 12 months old.
Delayed growth - head circumference | when the child is 24 months old.
  Head circumference in centimeters measured by a physical examination of the child when the child is 24 months old.
Knowledge of SIDS (sudden infant death syndrome) prevention | when the child is 6 months old.
  Knowledge of SIDS (sudden infant death syndrome) prevention as measured by the number of questions the mother answered correctly about SIDS prevention when the child is 6 months old. The questionnaire testing the mother's knowledge of SIDS is composed of five items from the Korean National Health Insurance Service's Infant Health Examination Questionnaire.
Vaccination | when the child is 6 months old.
  Vaccination as assessed by the completion of recommended vaccinations (tuberculosis, hepatitis B, Haemophilus influenzae type b (Hib), DTaP, polio, Streptococcus pneumoniae) when the child is 6 months old.
Vaccination | when the child is 12 months old.
  Vaccination as assessed by the completion of recommended vaccinations (tuberculosis, hepatitis B, Haemophilus influenzae type b (Hib), DTaP, polio, Streptococcus pneumoniae) when the child is 12 months old.
Vaccination | when the child is 24 months old.
  Vaccination as assessed by the completion of recommended vaccinations (tuberculosis, hepatitis B, Haemophilus influenzae type b (Hib), DTaP, polio, Streptococcus pneumoniae) when the child is 24 months old.
National health check-ups | when the child is 6 months old.
  National health check-ups assessed by asking whether the mother has visited a health center or pediatrician for an infant health checkup when the child is 6 months old.
National health check-ups | when the child is 12 months old.
  National health check-ups assessed by asking whether the mother has visited a health center or pediatrician for an infant health checkup when the child is 12 months old.
National health check-ups | when the child is 24 months old.
  National health check-ups assessed by asking whether the mother has visited a health center or pediatrician for an infant health checkup when the child is 24 months old.
Spousal participation in parenting | when the child is 6 months old.
  Spousal participation in parenting as measured by a questionnaire composed of 4 items when the child is 6 months old. The questionnaire was developed by Hong (1995) and used in the Panel Study on Korean Children (PSKC). The minimum score is 4 and the maximum score is 20, and a higher score means a better outcome.
Spousal participation in parenting | when the child is 12 months old.
  Spousal participation in parenting as measured by a questionnaire composed of 4 items when the child is 12 months old. The questionnaire was developed by Hong (1995) and used in the Panel Study on Korean Children (PSKC). The minimum score is 4 and the maximum score is 20, and a higher score means a better outcome.
Spousal participation in parenting | when the child is 24 months old.
  Spousal participation in parenting as measured by a questionnaire composed of 4 items when the child is 24 months old. The questionnaire was developed by Hong (1995) and used in the Panel Study on Korean Children (PSKC). The minimum score is 4 and the maximum score is 20, and a higher score means a better outcome.
Parenting related household expenses | when the child is 6 months old.
  Parenting-related household expenses, which measure a household's expenditures for pregnancy, childbirth, and supplies needed to care for the child when the child is 6 months old.
Parenting related household expenses | when the child is 12 months old.
  Parenting-related household expenses, which measure a household's expenditures for pregnancy, childbirth, and supplies needed to care for the child when the child is 12 months old.
Parenting related household expenses | when the child is 24 months old.
  Parenting-related household expenses, which measure a household's expenditures for pregnancy, childbirth, and supplies needed to care for the child when the child is 24 months old.
Intention to have another child | when the child is 24 months old.
  Intention to have another child as assessed by a single question, "Do you have any intention to have more children in the future?". Responses to this question are categorized into three options: "Yes, I have the intention to have another child", "No, I don't have the intention to have another child", and "I don't know."
Experience of delivery in the past 2 years | when the child is 24 months old.
  Experience of delivery in the past 2 years as assessed by using a single question: "Have you had the experience of subsequent childbirth (having another child after participating in the study) or are you currently pregnant?" Responses to this question are categorized into three options: "Yes, I have had subsequent childbirth experience," "Yes, I am currently pregnant," and "No, I don't have subsequent childbirth."
Depression (EPDS) | when the child is 6 months old.
  Depression as assessed using the EPDS (Edinburgh Postnatal Depression Scale) when the child is 6 months old. The EPDS (Edinburgh Postnatal Depression Scale) was developed by Cox et al. (1987) as a tool measuring postnatal depression. It is composed of 10 items. The minimum score is 0 and the maximum score is 30, and a higher score means a worse outcome.
Depression (EPDS) | when the child is 12 months old.
  Depression as assessed using the EPDS (Edinburgh Postnatal Depression Scale) when the child is 12 months old. The EPDS (Edinburgh Postnatal Depression Scale) was developed by Cox et al. (1987) as a tool measuring postnatal depression. It is composed of 10 items. The minimum score is 0 and the maximum score is 30, and a higher score means a worse outcome.
Depression (EPDS) | when the child is 24 months old.
  Depression as assessed using the EPDS (Edinburgh Postnatal Depression Scale) when the child is 24 months old. The EPDS (Edinburgh Postnatal Depression Scale) was developed by Cox et al. (1987) as a tool measuring postnatal depression. It is composed of 10 items. The minimum score is 0 and the maximum score is 30, and a higher score means a worse outcome.
Suicidal ideation | when the child is 6 months old.
  Suicidal ideation as assessed using the 10th item of EPDS (Edinburgh Postnatal Depression Scale) when the child is 6 months old. The EPDS (Edinburgh Postnatal Depression Scale) was developed by Cox et al. (1987) as a tool measuring postnatal depression and the 10th item of EPDS asks respondents to indicate how often they have experienced thoughts of self harm using a 4-point frequency scale.
Suicidal ideation | when the child is 12 months old.
  Suicidal ideation as assessed using the 10th item of EPDS (Edinburgh Postnatal Depression Scale) when the child is 12 months old. The EPDS (Edinburgh Postnatal Depression Scale) was developed by Cox et al. (1987) as a tool measuring postnatal depression and the 10th item of EPDS asks respondents to indicate how often they have experienced thoughts of self harm using a 4-point frequency scale.
Suicidal ideation | when the child is 24 months old.
  Suicidal ideation as assessed using the 10th item of EPDS (Edinburgh Postnatal Depression Scale) when the child is 24 months old. The EPDS (Edinburgh Postnatal Depression Scale) was developed by Cox et al. (1987) as a tool measuring postnatal depression and the 10th item of EPDS asks respondents to indicate how often they have experienced thoughts of self harm using a 4-point frequency scale.
Depression (PHQ-9) | when the child is 6 months old.
  Depression as assessed using the PHQ-9 (Patient Health Questionnaire-9) when the child is 6 months old. The PHQ-9 (Patient Health Questionnaire-9) was developed by Kroenke, K. et al. (2001) as a tool measuring the depression level of adults and composed of 9 items. The minimum score is 0 and the maximum score is 27, and higher score means a worse outcome.
Depression (PHQ-9) | when the child is 12 months old.
  Depression as assessed using the PHQ-9 (Patient Health Questionnaire-9) when the child is 12 months old. The PHQ-9 (Patient Health Questionnaire-9) was developed by Kroenke, K. et al. (2001) as a tool measuring the depression level of adults and composed of 9 items. The minimum score is 0 and the maximum score is 27, and higher score means a worse outcome.
Depression (PHQ-9) | when the child is 24 months old.
  Depression as assessed using the PHQ-9 (Patient Health Questionnaire-9) when the child is 24 months old. The PHQ-9 (Patient Health Questionnaire-9) was developed by Kroenke, K. et al. (2001) as a tool measuring the depression level of adults and composed of 9 items. The minimum score is 0 and the maximum score is 27, and higher score means a worse outcome.
Depression (Whooley & Arroll questions) | when the child is 6 weeks old.
  Maternal depression as assessed using the Whooley & Arroll questions when the child is 6 weeks old. To screen depression in outpatient settings, a simple tool called " two screening questions" was developed. Arroll B. et al. (2005) enhanced the sensitivity and specificity of the tool by adding a "help-seeking question". If the response to at least one of the Screening 2-Item questions is affirmative or if the response to the help-seeking question is affirmative, further evaluation is necessary.
Depression (Whooley & Arroll questions) | when the child is 18 months old.
  Maternal depression as assessed using the Whooley & Arroll questions when the child is 18 months old. To screen depression in outpatient settings, a simple tool called " two screening questions" was developed. Arroll B. et al. (2005) enhanced the sensitivity and specificity of the tool by adding a "help-seeking question". If the response to at least one of the Screening 2-Item questions is affirmative or if the response to the help-seeking question is affirmative, further evaluation is necessary.
Anxiety | when the child is 6 months old.
  Anxiety level as assessed using the GAD-2 (Generalized Anxiety Disorder 2-item) when the child is 6 months old. The GAD-2 (Generalized Anxiety Disorder 2-item) is a 2-item questionnaire that measures core anxiety symptoms. The minimum score is 0 and the maximum score is 6, and higher score means a worse outcome.
Anxiety | when the child is 12 months old.
  Anxiety level as assessed using the GAD-2 (Generalized Anxiety Disorder 2-item) when the child is 12 months old. The GAD-2 (Generalized Anxiety Disorder 2-item) is a 2-item questionnaire that measures core anxiety symptoms. The minimum score is 0 and the maximum score is 6, and higher score means a worse outcome.
Anxiety | when the child is 24 months old.
  Anxiety level as assessed using the GAD-2 (Generalized Anxiety Disorder 2-item) when the child is 24 months old. The GAD-2 (Generalized Anxiety Disorder 2-item) is a 2-item questionnaire that measures core anxiety symptoms. The minimum score is 0 and the maximum score is 6, and higher score means a worse outcome.
Maternal tobacco use | when the child is 6 months old.
  Maternal tobacco use assessed by current tobacco use status when the child is 6 months old. Maternal tobacco use is assessed by questioning the participants about their current tobacco use behavior during the month before the study.
Maternal tobacco use | when the child is 12 months old.
  Maternal tobacco use assessed by current tobacco use status when the child is 12 months old. Maternal tobacco use is assessed by questioning the participants about their current tobacco use behavior during the month before the study.
Maternal tobacco use | when the child is 24 months old.
  Maternal tobacco use assessed by current tobacco use status when the child is 24 months old. Maternal tobacco use is assessed by questioning the participants about their current tobacco use behavior during the month before the study.
Maternal alcohol consumption | when the child is 6 months old.
  Maternal alcohol consumption when the child is 6 months old. Maternal alcohol consumption is assessed by questioning the participants about their drinking behavior during the month before the study.
Maternal alcohol consumption | when the child is 12 months old.
  Maternal alcohol consumption when the child is 12 months old. Maternal alcohol consumption is assessed by questioning the participants about their drinking behavior during the month before the study.
Maternal alcohol consumption | when the child is 24 months old.
  Maternal alcohol consumption when the child is 24 months old. Maternal alcohol consumption is assessed by questioning the participants about their drinking behavior during the month before the study.
Delivery type | when the child is 6 weeks old.
  Delivery type as assessed by asking a mother to choose her delivery type between "normal delivery," "planned C-section," and "unplanned emergency C-section" when the child is 6 weeks old.
Maternal parenting stress | when the child is 6 months old.
  Maternal parenting stress as assessed using the Being a Mother Scale (BaM-13) when the child is 6 months old. The Being a Mother Scale (BaM-13) was developed by Matthey (2011) for assessing mothers' level of distress. It is composed of 13 items. The minimum score is 0 and the maximum score is 39, and a higher score means a high level of distress.
Maternal parenting stress | when the child is 12 months old.
  Maternal parenting stress as assessed using the Being a Mother Scale (BaM-13) when the child is 12 months old. The Being a Mother Scale (BaM-13) was developed by Matthey (2011) for assessing mothers' level of distress. It is composed of 13 items. The minimum score is 0 and the maximum score is 39, and a higher score means a high level of distress.
Maternal parenting stress | when the child is 24 months old.
  Maternal parenting stress as assessed using the Being a Mother Scale (BaM-13) when the child is 24 months old. The Being a Mother Scale (BaM-13) was developed by Matthey (2011) for assessing mothers' level of distress. It is composed of 13 items. The minimum score is 0 and the maximum score is 39, and a higher score means a high level of distress.
Intimate partner violence | when the child is 6 months old.
  Intimate partner violence as assessed using the HITS (Hurt, Insult, Threaten, and Scream) tool when the child is 6 months old. The HITS (Hurt, Insult, Threaten, and Scream) tool was developed by Sherin et al. (1998) for assessing the level of domestic violence. It is composed of 4 items. The minimum score is 4 and the maximum score is 20, and higher score means a high level of domestic violence.
Intimate partner violence | when the child is 12 months old.
  Intimate partner violence as assessed using the HITS (Hurt, Insult, Threaten, and Scream) tool when the child is 12 months old. The HITS (Hurt, Insult, Threaten, and Scream) tool was developed by Sherin et al. (1998) for assessing the level of domestic violence. It is composed of 4 items. The minimum score is 4 and the maximum score is 20, and higher score means a high level of domestic violence.
Intimate partner violence | when the child is 24 months old.
  Intimate partner violence as assessed using the HITS (Hurt, Insult, Threaten, and Scream) tool when the child is 24 months old. The HITS (Hurt, Insult, Threaten, and Scream) tool was developed by Sherin et al. (1998) for assessing the level of domestic violence. It is composed of 4 items. The minimum score is 4 and the maximum score is 20, and higher score means a high level of domestic violence.
Maternal body weight | when the child is 6 weeks old.
  Maternal body weight when the child is 6 weeks old.
Maternal body weight | when the child is 6 months old.
  Maternal body weight when the child is 6 months old.
Maternal body weight | when the child is 12 months old.
  Maternal body weight when the child is 12 months old.
Maternal body weight | when the child is 24 months old.
  Maternal body weight when the child is 24 months old.
Social support | when the child is 6 months old.
  Social support as measured by a questionnaire developed by the Korea Institute of Child Care and Education when the child is 6 months old. The questionnaire measuring social support developed and used by Korea Institute of Child Care and Education is composed of 12 items. The minimum score is 12 and the maximum score is 60, and a higher score means a better outcome.
Social support | when the child is 12 months old.
  Social support as measured by a questionnaire developed by the Korea Institute of Child Care and Education when the child is 12 months old. The questionnaire measuring social support developed and used by Korea Institute of Child Care and Education is composed of 12 items. The minimum score is 12 and the maximum score is 60, and a higher score means a better outcome.
Social support | when the child is 24 months old.
  Social support as measured by a questionnaire developed by the Korea Institute of Child Care and Education when the child is 24 months old. The questionnaire measuring social support developed and used by Korea Institute of Child Care and Education is composed of 12 items. The minimum score is 12 and the maximum score is 60, and a higher score means a better outcome.
Food insecurity | when the child is 12 months old.
  Food insecurity assessed by asking about the family's level of limited access to adequate food over the past year when the child is 12 months.
Food insecurity | when the child is 24 months old.
  Food insecurity assessed by asking about the family's level of limited access to adequate food over the past year when the child is 24 months.
Spousal intimacy | when the child is 6 months old.
  Spousal intimacy as measured using the Revised-Kansas Marital Satisfaction Scale modified by the Korea Institute of Child Care and Education when the child is 6 months old. The Revised-Kansas Marital Satisfaction Scale modified by the Korea Institute of Child Care and Education is composed of 4 items. The minimum score is 4 and the maximum score is 20, and higher score means a better outcome.
Spousal intimacy | when the child is 12 months old.
  Spousal intimacy as measured using the Revised-Kansas Marital Satisfaction Scale modified by the Korea Institute of Child Care and Education when the child is 12 months old. The Revised-Kansas Marital Satisfaction Scale modified by the Korea Institute of Child Care and Education is composed of 4 items. The minimum score is 4 and the maximum score is 20, and higher score means a better outcome.
Spousal intimacy | when the child is 24 months old.
  Spousal intimacy as measured using the Revised-Kansas Marital Satisfaction Scale modified by the Korea Institute of Child Care and Education when the child is 24 months old. The Revised-Kansas Marital Satisfaction Scale modified by the Korea Institute of Child Care and Education is composed of 4 items. The minimum score is 4 and the maximum score is 20, and higher score means a better outcome.
Spousal tobacco use | when the child is 6 months old.
  Spousal tobacco use assessed by current tobacco use status when the child is 6 months old. Spouse tobacco use is assessed by questioning participants about their spouse's current tobacco use behavior during the month before the study.
Spousal tobacco use | when the child is 12 months old.
  Spousal tobacco use assessed by current tobacco use status when the child is 12 months old. Spouse tobacco use is assessed by questioning participants about their spouse's current tobacco use behavior during the month before the study.
Spousal tobacco use | when the child is 24 months old.
  Spousal tobacco use assessed by current tobacco use status when the child is 24 months old. Spouse tobacco use is assessed by questioning participants about their spouse's current tobacco use behavior during the month before the study.
Spousal alcohol consumption | when the child is 6 months old.
  Spousal alcohol consumption when the child is 6 months old. Spouse alcohol consumption is assessed by questioning participants about their spouse's drinking behavior during the month before the study.
Spousal alcohol consumption | when the child is 12 months old.
  Spousal alcohol consumption when the child is 12 months old. Spouse alcohol consumption is assessed by questioning participants about their spouse's drinking behavior during the month before the study.
Spousal alcohol consumption | when the child is 24 months old.
  Spousal alcohol consumption when the child is 24 months old. Spouse alcohol consumption is assessed by questioning participants about their spouse's drinking behavior during the month before the study.
Parent-child interaction | when the child is 12 months old.
  Parent-child interaction as assessed by using the NCAST (Nursing Child Assessment Teaching Scale) when the child is 12 months old. The NCAST (Nursing Child Assessment Teaching Scale) was developed by Barnard (1989) for assessing parent-child interaction. It is composed of 73 items that measure sensitivity to cues, response to child's distress, cognitive growth fostering, clarity of cues, and responsiveness to caregiver. The minimum score is 0 and the maximum score is 105, and a higher score means a better outcome.
Parent-child interaction | when the child is 24 months old.
  Parent-child interaction as assessed by using the NCAST (Nursing Child Assessment Teaching Scale) when the child is 24 months old. The NCAST (Nursing Child Assessment Teaching Scale) was developed by Barnard (1989) for assessing parent-child interaction. It is composed of 73 items that measure sensitivity to cues, response to child's distress, cognitive growth fostering, clarity of cues, and responsiveness to caregiver. The minimum score is 0 and the maximum score is 105, and a higher score means a better outcome.
Safety knowledge | when the child is 42 months old
  Maternal safety knowledge assessed through age-appropriate questionnaire items from the Korean National Health Insurance Service's child Health Examination Questionnaire when the child is 42 months old.
Safety knowledge | when the child is 54 months old
  Maternal safety knowledge assessed through age-appropriate questionnaire items from the Korean National Health Insurance Service's child Health Examination Questionnaire when the child is 54 months old.
Safety knowledge | when the child is 66 months old
  Maternal safety knowledge assessed through age-appropriate questionnaire items from the Korean National Health Insurance Service's child Health Examination Questionnaire when the child is 66 months old.
Emergency department visits due to injuries (maternal-report) | when the child is 42 months old.
  Number of emergency department visits due to injuries as reported by mothers when the child is 42 months old.
Emergency department visits due to injuries (maternal-report) | when the child is 54 months old.
  Number of emergency department visits due to injuries as reported by mothers when the child is 54 months old.
Emergency department visits due to injuries (maternal-report) | when the child is 66 months old.
  Number of emergency department visits due to injuries as reported by mothers when the child is 66 months old.
Hospital admission (maternal-report) | when the child is 66 months old.
  Number of hospital admission as reported by mothers when the child is 66 months old.
Spousal participation in parenting | when the child is 66 months old.
  Spousal participation in parenting as measured by a questionnaire composed of 4 items when the child is 66 months old. The questionnaire was developed by Hong (1995) and used in the Panel Study on Korean Children (PSKC). The minimum score is 4 and the maximum score is 20, and a higher score means a better outcome.
Parenting related household expenses | when the child is 66 months old.
  Parenting-related household expenses, which measure a household's expenditures for pregnancy, childbirth, and supplies needed to care for the child when the child is 66 months old.
Subsequent childbirth after study participation | when the child is 66 months old.
  Experience of subsequent childbirth after study participation as assessed by using a single question: "Have you had the experience of subsequent childbirth (having another child after participating in the study) or are you currently pregnant?" Responses to this question are categorized into three options: "Yes, I have had subsequent childbirth experience," "Yes, I am currently pregnant," and "No, I don't have subsequent childbirth."
Anxiety | when the child is 42 months old.
  Maternal anxiety level as assessed using the GAD-2 (Generalized Anxiety Disorder 2-item) scale when the child is 42 months old. The GAD-2 has a score range of 0-6, with higher scores indicating greater anxiety levels.
Anxiety | when the child is 54 months old.
  Maternal anxiety level as assessed using the GAD-2 (Generalized Anxiety Disorder 2-item) scale when the child is 54 months old. The GAD-2 has a score range of 0-6, with higher scores indicating greater anxiety levels.
Anxiety | when the child is 66 months old.
  Maternal anxiety level as assessed using the GAD-7 (Generalized Anxiety Disorder 7-item) scale when the child is 66 months old. The GAD-7 has a score range of 0-21, with higher scores indicating greater anxiety levels.
Maternal tobacco use | when the child is 66 months old.
  Maternal tobacco use assessed by current tobacco use status when the child is 66 months old. Maternal tobacco use is assessed by questioning the participants about their current tobacco use behavior during the month before the study.
Maternal alcohol consumption | when the child is 66 months old.
  Maternal alcohol consumption when the child is 66 months old. Maternal alcohol consumption is assessed by questioning the participants about their drinking behavior during the month before the study.
Maternal parenting stress | when the child is 66 months old.
  Maternal parenting stress as assessed using a questionnaire when the child is 66 months old. The questionnaire will measure maternal stress associated with parenting roles and childcare responsibilities, with higher scores indicating greater levels of parenting-related stress.
Intimate partner violence | when the child is 66 months old.
  Intimate partner violence as assessed using the HITS (Hurt, Insult, Threaten, and Scream) tool when the child is 66 months old. The HITS (Hurt, Insult, Threaten, and Scream) tool was developed by Sherin et al. (1998) for assessing the level of domestic violence. It is composed of 4 items. The minimum score is 4 and the maximum score is 20, and higher score means a high level of domestic violence.
Social support | when the child is 66 months old.
  Social support as measured by a questionnaire developed by the Korea Institute of Child Care and Education when the child is 66 months old. The questionnaire is composed of 12 items. The minimum score is 12 and the maximum score is 60, and a higher score means a better outcome.
Food insecurity | when the child is 66 months old.
  Food insecurity assessed by asking about the family's level of limited access to adequate food over the past year when the child is 66 months.
Spousal intimacy | when the child is 66 months old.
  Spousal intimacy as measured using the Revised-Kansas Marital Satisfaction Scale modified by the Korea Institute of Child Care and Education when the child is 66 months old. The Scale is composed of 4 items. The minimum score is 4 and the maximum score is 20, and higher score means a better outcome.
Spousal tobacco use | when the child is 66 months old.
  Spousal tobacco use assessed by current tobacco use status when the child is 66 months old. Spouse tobacco use is assessed by questioning participants about their spouse's current tobacco use behavior during the month before the study.
Spousal alcohol consumption | when the child is 66 months old.
  Spousal alcohol consumption when the child is 66 months old. Spouse alcohol consumption is assessed by questioning participants about their spouse's drinking behavior during the month before the study.
Maternal employment status | when the child is 42 months old.
  Maternal employment status as assessed via self-report questionnaire when the child is 42 months old. Employment status will be categorized as employed (returned to pre-birth job, new employment, on leave), attending school, or unemployed/not in school using a simplified questionnaire adapted from the Korea Early Childhood Education and Care Panel Study.
Maternal employment status | when the child is 54 months old.
  Maternal employment status as assessed via self-report questionnaire when the child is 54 months old. Employment status will be categorized as employed (returned to pre-birth job, new employment, on leave), attending school, or unemployed/not in school using a simplified questionnaire adapted from the Korea Early Childhood Education and Care Panel Study.
Maternal employment status | when the child is 66 months old.
  Maternal employment status as assessed via self-report questionnaire when the child is 66 months old. A comprehensive questionnaire adapted from the Panel Study on Korean Children will be used to collect detailed information, including specific occupation type and workplace position.
Paternal employment status (maternal-report) | when the child is 66 months old
  Father's employment status will be assessed through maternal-report questionnaire adapted from the Panel Study on Korean Children when the child is 66 months old.
Monthly household income | when the child is 66 months old
  Self-reported average monthly household income over the past 12 months, measured in Korean Won.
Basic livelihood security status | when the child is 66 months old.
  Household classification under the National Basic Livelihood Security Act, categorized as basic livelihood security recipient, near-poor household, not applicable, or unknown.
Maternal marital status | when the child is 42 months old.
  Mother's marital status changes over time, categorized as single, married (first marriage), married (remarried), widowed, divorced, or separated when the child is 42 months old.
Maternal marital status | when the child is 54 months old.
  Mother's marital status changes over time, categorized as single, married (first marriage), married (remarried), widowed, divorced, or separated when the child is 54 months old.
Maternal marital status | when the child is 66 months old.
  Mother's marital status changes over time, categorized as single, married (first marriage), married (remarried), widowed, divorced, or separated when the child is 66 months old.
Child's Educational facility attendance | when the child is 42 months old.
  Self-reported enrollment status and type of educational facility currently attended by the child when the child is 42 months old.
Child's Educational facility attendance | when the child is 54 months old.
  Self-reported enrollment status and type of educational facility currently attended by the child when the child is 54 months old.
Child's Educational facility attendance | when the child is 66 months old.
  Self-reported enrollment status and type of educational facility currently attended by the child when the child is 66 months old.
Parental efficacy | when the child is 42 months old.
  Parental efficacy as assessed using a modified version of the Parenting Sense of Competence Scale originally developed by Gibaud-Wallston & Wandersman (1978) when the child is 42 months old. The instrument consists of 16 items rated on a 5-point scale.
Parental efficacy | when the child is 54 months old.
  Parental efficacy as assessed using a modified version of the Parenting Sense of Competence Scale originally developed by Gibaud-Wallston & Wandersman (1978) when the child is 54 months old. The instrument consists of 16 items rated on a 5-point scale.
Parental efficacy | when the child is 66 months old.
  Parental efficacy as assessed using a modified version of the Parenting Sense of Competence Scale originally developed by Gibaud-Wallston & Wandersman (1978) when the child is 66 months old. The instrument consists of 16 items rated on a 5-point scale.
Self-efficacy | when the child is 66 months old.
  Self-efficacy as assessed using the Self-Efficacy Scale originally developed by Pearlin et al. (1981). The Korean version was adapted by the Korea Institute of Child Care and Education and consists of 4 items rated on a 5-point Likert scale.
Healthcare utilization (administrative data) | when the child is 66 months old.
  Number of outpatient visits and number of hospital admissions obtained through linkage with National Health Insurance Service data.
National health check-ups (administrative data) | when the child is 66 months old.
  Participation in national health screening programs obtained through linkage with National Health Insurance Service data when the child is 66 months old.
Child lifestyle habits | when the child is 66 months old.
  Child lifestyle habits as assessed using selected items appropriate for 66-month-old children. The original tool was developed by Allen & Martoz (2003, 2007) and adapted and validated by the Panel Study on Korean Children (PSKC) research team. The assessment includes: (1) Daily sleep duration measured in hours, (2) Meal time regularity rated on a 5-point scale, (3) Weekly breakfast frequency at home, and (4) Media use frequency and age of first use for digital devices rated on a 5-point scale.
Child problem behavior | when the child is 66 months old.
  Child problem behavior as assessed using 10 items translated from the problem behavior section of the Korean version of Social Skills Rating System for preschool level (K-SSRS).
Child social-emotional development (social competence) | when the child is 66 months old.
  Child's social-emotional development as assessed using the social skills section of the Korean version of Social Skills Rating System for preschool level (K-SSRS). The instrument consists of 32 items originally used in the Panel Study on Korean Children (PSKC).
Child BMI | when the child is 66 months old.
  BMI calculated from height and weight measurements (kg/m²) obtained through physical examination.
Child dental caries | when the child is 66 months old.
  Dental caries screening using the "lift the lip" screening method to assess tooth decay.
Child health status | when the child is 42 months old.
  Mother's perception of her child's overall health status rated on a 5-point scale when the child is 42 months old.
Child health status | when the child is 54 months old.
  Mother's perception of her child's overall health status rated on a 5-point scale when the child is 54 months old.
Child health status | when the child is 66 months old.
  Mother's perception of her child's overall health status rated on a 5-point scale when the child is 66 months old.
Maternal self-rated health | when the child is 42 months old.
  Mother's perception of her own health status rated on a 5-point scale when the child is 42 months old.
Maternal self-rated health | when the child is 54 months old.
  Mother's perception of her own health status rated on a 5-point scale when the child is 54 months old.
Maternal self-rated health | when the child is 66 months old.
  Mother's perception of her own health status rated on a 5-point scale when the child is 66 months old.
Vaccination (administrative data) | when the child is 66 months old.
  Vaccination completion information obtained through linkage with Korea Disease Control and Prevention Agency vaccination data.
Community service linkage | when the child is 66 months old.
  Community service linkage as measured by the number of community services a mother has received during the last year.
Maternal quality of life | when the child is 66 months old.
  Mother's overall quality of life assessed through self-report questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ho Khang, MD, PhD, Principal Investigator — Seoul National University College of Medicine
Locations (2):
- South Korea (2):
  - Institute of Health Policy and Management, Medical Research Center, Seoul National University, Seoul
  - Medical Research Collaborating Center, Seoul National University Biomedical Research Institute, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khang YH, Kim YM, Kim JH, Yu J, Oh R, June KJ, Cho SH, Lee JY, Cho HJ. Impact of the Korea Early Childhood Home-visiting Intervention (KECHI) on child health and development and maternal health: a randomised controlled trial protocol. BMJ Open. 2024 Aug 8;14(8):e082434. doi: 10.1136/bmjopen-2023-082434. PMID 39122404
- [Background] June KJ, Lee JY, Cho SH. Infant Mother's Experiences with the Sustained Nurse Home-Visiting Program. J Korean Soc Matern Child Health. 2021;25(1):31-41.
- [Background] Khang YH, Cho SH, June KJ, Lee JY, Kim YM, Cho HJ. The Seoul healthy first step project: Introduction and expansion, program content and performance, and future challenges. Journal of the Korean Society of Maternal and Child Health. 2018;22(2):63-76.
- [Background] Lee JY, June KJ, Cho S-H. Competencies of nurses in a maternal early childhood sustained home-visiting program. Journal of Korean Academy of Community Health Nursing. 2017;28(4):397-409.